CLINICAL TRIAL: NCT00845520
Title: A Prospective Multi-center Clinical Study to Evaluate the Safety and Effectiveness of the Light Adjustable Lens (LAL) in Subjects Undergoing Cataract Extraction
Brief Title: Safety and Effectiveness of the Calhoun Vision Light Adjustable Intraocular Lens (LAL)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Calhoun Vision, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSP 002-00
Record Dates: First submitted 2009-02-13; First posted 2009-02-18 (Estimated); Results first posted 2018-07-06 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2018-06

CONDITIONS: Cataracts
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Intervention Model Description: Phase 2 medical device study
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lens implantation +1.00 diopter (D) postop target (Experimental): Lens implant power calculated for postoperative MRSE target of +1.00 D
  Interventions: Device: Lens implantation +1.00 D postop target
- Lens implantation -1.00 D postop target (Experimental): Lens implant power calculated for postoperative MRSE target of -1.00 D
  Interventions: Device: Lens implantation -1.00 D postop target
- Lens implantation 0.00 D postop target (Experimental): Lens implant power calculated for postoperative MRSE target of 0.00 D
  Interventions: Device: Lens implantation 0.00 D postop target

INTERVENTIONS:
Device: Lens implantation +1.00 D postop target — Lens implantation +1.00 D postoperative MRSE target. Light Delivery Device treatment based on postoperative manifest refraction.
  Other Names: Light Delivery Device
  Arms: Lens implantation +1.00 diopter (D) postop target
Device: Lens implantation -1.00 D postop target — Lens implantation -1.00 D postoperative MRSE target. Light Delivery Device treatment based on postoperative manifest refraction.
  Other Names: Light Delivery Device
  Arms: Lens implantation -1.00 D postop target
Device: Lens implantation 0.00 D postop target — Lens implantation 0.00 D postoperative MRSE target. Light Delivery Device treatment based on postoperative manifest refraction.
  Other Names: Light Delivery Device
  Arms: Lens implantation 0.00 D postop target

SUMMARY:
The primary objective of this study is to evaluate, for the visual correction of aphakia, the safety and effectiveness of the Calhoun Vision Light Adjustable intraocular lens (LAL) and Light Delivery Device (LDD) in treating postoperative residual refractive error by providing a stable, targeted refractive adjustment of the LAL power and lock-in treatments with the LDD.

ELIGIBILITY:
Inclusion Criteria:

* Pre-operative regular corneal astigmatism less than or equal to 1.00 diopters by keratometry.
* Adults between the ages of 40 and 80 inclusive.
* Cataract causing reduction in best spectacle-corrected visual acuity to a level of 20/32 or worse.
* Best corrected visual acuity projected (by clinical estimate based upon past ocular history and retinal exam) to be 20/25 or better after cataract removal and IOL implantation.
* Clear intraocular media other than cataract.
* Potentially good vision in the fellow eye with BCVA 20/40 or better.
* Willing and able to comply with the schedule for power adjustment/lock-in treatments and the schedule for follow-up visits.
* Fully dilated pupil diameter of more than or equal to 7.0 mm.

Exclusion Criteria:

* Zonular laxity or dehiscence.
* Pseudoexfoliation.
* Age related macular degeneration involving the presence of geographic atrophy or soft drusen.
* Retinal degenerative disorder that is expected to cause future vision loss.
* Diabetes with any evidence of retinopathy.
* Evidence of glaucomatous optic neuropathy.
* History of uveitis.
* Significant anterior segment pathology, such as rubeosis iridis, aniridia, or iris coloboma.
* Corneal pathology that is either progressive or sufficient to reduce BCVA to 20/25 or worse.
* Keratoconus or suspected of having keratoconus.
* Corneal dystrophy including basement membrane dystrophy.
* Previous corneal or intraocular surgery
* Systemic medication that may increase sensitivity to UV light such as tetracycline, doxycycline, psoralens, amiodarone, and phenothiazines.
* Complications during cataract surgery including posterior capsule rupture, zonular rupture, radial capsulorhexis tear, vitreous loss, iris trauma, corneal complications or any intraoperative abnormality that may affect the postoperative pupillary dilation, or the centration or tilt of the intraocular lens.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2009-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: R. Doyle Stulting, MD, PhD, Principal Investigator — Emory Eye Center
Locations (6):
- United States (5):
  - Altos Eye Physicians, Los Altos, California
  - Maloney Vision Institute, Los Angeles, California
  - Price Vision Group, Indianapolis, Indiana
  - Discover Vision Centers, Leawood, Kansas
  - Pepose Vision Institute, Chesterfield, Missouri
- CODET Vision Institute, Tijuana, Zona Rio, Mexico

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: eyes
Groups:
- Lens Implant Power +1.00 D Target: Lens implant power +1.00 D target: Subjects who require cataract extraction and intraocular lens implantation are implanted with the Light Adjustable Lens with a postoperative +1.00 D MRSE target. At 17 to 21 days, the manifest refraction is measured and the implanted LAL is treated with a targeted dose of light using the Light Delivery Device to produce a modification in the lens curvature, resulting in a predictable change in refractive power.
- Lens Implant Power -1.00 D Target: Lens implant power -1.00 D target: Subjects who require cataract extraction and intraocular lens implantation are implanted with the Light Adjustable Lens with a postoperative -1.00 D MRSE target. At 17 to 21 days, the manifest refraction is measured and the implanted LAL is treated with a targeted dose of light using the Light Delivery Device to produce a modification in the lens curvature, resulting in a predictable change in refractive power.
- Lens Implant Power 0.00 D Target: Lens implant power 0.00 D target: Subjects who require cataract extraction and intraocular lens implantation are implanted with the Light Adjustable Lens with a postoperative 0.00 D MRSE target. At 17 to 21 days, the manifest refraction is measured and the implanted LAL is treated with a targeted dose of light using the Light Delivery Device to produce a modification in the lens curvature, resulting in a predictable change in refractive power.
Period: Overall Study
Arm/Group | Lens Implant Power +1.00 D Target | Lens Implant Power -1.00 D Target | Lens Implant Power 0.00 D Target
Started | 25; 25 eyes | 25; 25 eyes | 24; 24 eyes
Completed | 23; 23 eyes | 23; 23 eyes | 23; 23 eyes
Not Completed | 2; 2 eyes | 2; 2 eyes | 1; 1 eyes
Not completed — Death | 1 | 2 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Lens Implant Power +1.00 D Target: The eyes would have a post-surgical Manifest Refraction Spherical Equivalent (MRSE) target of +1.00 diopter
- Lens Implant Power 0.00 D Target: The eyes would have a post-surgical Manifest Refraction Spherical Equivalent (MRSE) target of 0.00 diopter
- Lens Implant Power -1.00 D Target: The eyes would have a post-surgical Manifest Refraction Spherical Equivalent (MRSE) target of 11.00 diopter
- Total: Total of all reporting groups
Arm/Group | Lens Implant Power +1.00 D Target | Lens Implant Power 0.00 D Target | Lens Implant Power -1.00 D Target | Total
Number analyzed (Participants) | 25 | 24 | 25 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.3 (9.3) | 65.6 (7.3) | 65.9 (9.2) | 66.1 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 17 | 12 | 44
  Male | 10 | 7 | 13 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 21 | 15 | 19 | 55
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 8 | 6 | 17

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Eyes Achieving a Manifest Refraction Spherical Equivalent (MRSE) Within ± 0.50 D of the Intended Adjustment Target
Description: Predictability of post-operative refractive adjustments of the implanted LAL, with 75% of the eyes achieving a manifest refraction spherical equivalent (MRSE) within ± 0.50 D of the intended adjustment target at the point of stability. All three arms of the study had the same end point so the results were presented as one combined cohort.
Time Frame: 6 months post-operative
Population: ITT
Measure: Number; unit: percentage of eyes
Groups:
- Lens Implant Power -1.00 D Target: Eyes randomized to a target lens implant power of -1.00 D
- Lens Implant Power +1.00 D Target: Eyes randomized to a target lens implant power of +1.00 D
- Lens Implant Power 0.00 D Target: Eyes randomized to a target lens implant power of 0.00 D
Arm/Group | Lens Implant Power -1.00 D Target | Lens Implant Power +1.00 D Target | Lens Implant Power 0.00 D Target
Number analyzed (Participants) | 23 | 25 | 24
percentage of eyes | 78.3 | 80.0 | 79.2

2. Secondary Outcome: Percentage of Participants With Eyes With Improvement in Uncorrected Visual Acuity (UCVA)
Description: Improvement in uncorrected visual acuity (UCVA): For those best case eyes with a pre-light treatment UCVA of 20/50 or worse, 65% of eyes should have an uncorrected visual acuity of 20/40 or better at the refractive stable point after the adjustment and lock-in treatments. All three arms of the study had the same end point so the results were presented as one combined cohort.
Time Frame: 6 months post operative
Population: Participants with eyes with UCVA of 20/50 or worse UCVA prior to light treatment
Measure: Number; unit: percentage of eyes
Groups:
- Lens Implant Power -1.00 D Target: Eyes randomized to a target of -1.00 D
- Lens Implant Power of +1.00 D: Eyes randomized to a target of +1.00 D
- Lens Implant Power of 0.0 D Target: Eyes randomized to a target of 0.0 D
Arm/Group | Lens Implant Power -1.00 D Target | Lens Implant Power of +1.00 D | Lens Implant Power of 0.0 D Target
Number analyzed (Participants) | 10 | 1 | 1
percentage of eyes | 77.8 | 100 | 0

3. Other Pre Specified Outcome: Percentage of Eyes With Best Corrected Visual Acuity (BSCVA) of 20/40 or Better
Description: Best Corrected Visual Acuity (BSCVA): The percentage of eyes achieving overall and best case BSCVA of 20/40 or better should be comparable to the FDA grid of historical controls for intraocular lenses. All three arms of the study had the same end point so the results were presented as one combined cohort.
Time Frame: 12 months
Population: All available eyes at 12 months. The overall number of participants for this outcome measures differs the previously stated overall number of 74 because two subjects were deceased at their 12 month post-operative follow up visit.
Measure: Number; unit: percentage of eyes
Groups:
- Lens Implant Power With -1.00 D Target: Eyes randomized to a postoperative target MRSE of -1.00 D
- Lens Implant Power With 0.00 D Target: Eyes randomized to a postoperative target MRSE of 0.00 D
- Lens Implant Power With +1.00 D Target: Eyes randomized to a postoperative target MRSE of +1.00 D
Arm/Group | Lens Implant Power With -1.00 D Target | Lens Implant Power With 0.00 D Target | Lens Implant Power With +1.00 D Target
Number analyzed (Participants) | 23 | 24 | 25
percentage of eyes | 100 | 100 | 100

ADVERSE EVENTS:
Time Frame: 36 months
Groups:
- Lens Implant Power of +1.00 D Target: Eyes with a post-surgical Manifest Refraction Spherical Equivalent (MRSE) target of +1.00 D
- Lens Implant Power of -1.00 D Target: Eyes with a post-surgical Manifest Refraction Spherical Equivalent (MRSE) target of -1.00 D
- Lens Implant Power of 0.00 D: Eyes with a post-surgical Manifest Refraction Spherical Equivalent (MRSE) target of 0.00 D
Arm/Group | Lens Implant Power of +1.00 D Target | Lens Implant Power of -1.00 D Target | Lens Implant Power of 0.00 D
All-Cause Mortality (participants affected / at risk) | 0/25 | 2/25 | 1/24
Serious Adverse Events (participants affected / at risk) | 3/25 | 2/25 | 1/24
Other Adverse Events (participants affected / at risk) | 18/25 | 15/25 | 14/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lens Implant Power of +1.00 D Target (N=25) | Lens Implant Power of -1.00 D Target (N=25) | Lens Implant Power of 0.00 D (N=24)
Secondary Surgical Intervention (Eye disorders) | 1 (1) | 1 (1) | 1 (1)
Stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Optic neuritis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
epiretinal membrane and macular hole (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
wet age related macular degeneration (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
macular edema secondary to epiretinal membrate (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
heart attack with pacemaker implanted (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lens Implant Power of +1.00 D Target (N=25) | Lens Implant Power of -1.00 D Target (N=25) | Lens Implant Power of 0.00 D (N=24)
Posterior Capsular Opacity (Eye disorders) | 17 (33) | 15 (37) | 13 (30)
Blepharitis (Eye disorders) | 1 (3) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No